CLINICAL TRIAL: NCT01340313
Title: Ultrasonographic Evaluation of Drug Spread in Epidural Space During Caudal Block in Children
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2010-0775
Record Dates: First submitted 2011-04-05; First posted 2011-04-22 (Estimated); Last update posted 2013-03-06 (Estimated); Status verified 2013-03

CONDITIONS: Children Who Need Urological Surgery
Keywords: caudal block, children, ultrasound, urological surgery

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1: 4 times evaluation according to doses in 1 group

SUMMARY:
Caudal block is the world-widely used technique for an effective postoperative analgesia in children undergoing OPD-based infra-umbilical surgery. Because the caudal block is usually performed with a single-shot, proper dosage is required to achieve sufficient analgesic levels. Several clinical researches have been performed to assess the drug spread levels using mathematical equation, X-ray evaluation, and ultrasonography during caudal block in children. In our previous study using fluoroscopy, we obtained the results that the established weight-based doses provided adequate block levels for each type of surgery.

Ultrasonography is precise tool to evaluate the spinal structures and can provide estimated information in real time during caudal or epidural block in children.

The aim of this study is to evaluate the drug spread level with a weight-based doses using ultrasonography during caudal block in children and assess the reliability of the real time ultrasonography to determine the drug spread levels. After general anesthesia, the patient will be placed in lateral decubitus position for caudal block. Total 1.5 ml/kg of 0.15% ropivacaine will be injected into the caudal space. The spread level will be step-wise evaluated using ultrasonography at the injected drug dose of 0.5 ml/kg, 1.0 ml/kg, 1.25 ml/kg, and 1.5 ml/kg.

ELIGIBILITY:
Inclusion Criteria:

* children who needed caudal block for postoperative analgesia (age 3 months ~ 5 years old)
* Consent from one of parents 3. ASA physical status I or II

Exclusion Criteria:

* bleeding tendency
* spinal anomaly
* infection focus on back
* allergic reaction to local anesthetics
* foreigner of illiteracy who cannot read consent form

Ages: 3 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: 3 months old ~ 5 years old children undergoing minor infra-umbilical urological surgery
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2011-03; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
drug spread level with a weight-based doses | every 10 seconds for 1 minute during drug injection (10, 20, 30, 40, 50, and 60 seconds).
  1. spread levels of drug within the epidural space during drug injection with caudal block at every doses using real-time ultrasound examination.
  2. maximum spread levels within the epidural space

CONTACTS AND LOCATIONS:
Overall Officials: Hae Kum Kil, MD, MS, Principal Investigator — Severance Hospital
Locations (1):
- Hae Keum Kil, Seoul, Seoul, South Korea

REFERENCES:
- [Background] Hong JY, Han SW, Kim WO, Cho JS, Kil HK. A comparison of high volume/low concentration and low volume/high concentration ropivacaine in caudal analgesia for pediatric orchiopexy. Anesth Analg. 2009 Oct;109(4):1073-8. doi: 10.1213/ane.0b013e3181b20c52. PMID 19762734
- [Background] Shin SK, Hong JY, Kim WO, Koo BN, Kim JE, Kil HK. Ultrasound evaluation of the sacral area and comparison of sacral interspinous and hiatal approach for caudal block in children. Anesthesiology. 2009 Nov;111(5):1135-40. doi: 10.1097/ALN.0b013e3181bc6dd4. PMID 19809281
- [Background] Koo BN, Hong JY, Kil HK. Spread of ropivacaine by a weight-based formula in a pediatric caudal block: a fluoroscopic examination. Acta Anaesthesiol Scand. 2010 May;54(5):562-5. doi: 10.1111/j.1399-6576.2010.02224.x. Epub 2010 Mar 10. PMID 20236099
- [Background] Lundblad M, Lonnqvist PA, Eksborg S, Marhofer P. Segmental distribution of high-volume caudal anesthesia in neonates, infants, and toddlers as assessed by ultrasonography. Paediatr Anaesth. 2011 Feb;21(2):121-7. doi: 10.1111/j.1460-9592.2010.03485.x. Epub 2010 Dec 15. PMID 21159024